CLINICAL TRIAL: NCT06133088
Title: Explore the Efficacy and Safety of Dalpiciclib Combined With Fluvestrant and Compound Gossypol Acetate Tablets in Advanced HR-positive and HER2-negative Breast Cancer After CDK4/6 Treatment Failed.
Brief Title: Dalpiciclib Combination With Fulvestrant and Compound Gossyfol Acetate Tablets in Women With CDK4/6 Inhibitor-refractory HR-positive HER-2 Negtive Metastatic Breast Cancer: a Phase 2 Clinical Trial.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shao Xiying, Medical team leader, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIM-B002a
Record Dates: First submitted 2023-10-31; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Advanced HR-positive and HER2-negative Breast Cancer; CDK4/6 Inhibitor Treatment Failed
MeSH Terms: interventions — dalpiciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): This is a single-arm, Phase II clinical study to explore the efficacy and safety of dalpiciclib combined with fluvestrant and compound gossypol acetate tablets in advanced HR-positive and HER2-negative breast cancer after CDK4/6 treatment failed.
  Interventions: Drug: dalpiciclib; fluvestrant; compound gossypol acetate tablets

INTERVENTIONS:
Drug: dalpiciclib; fluvestrant; compound gossypol acetate tablets — Darcilie: 150mg orally for three weeks and stop for one week. Fluvestrant: 500mg every four weeks. A further 500mg dose two weeks after the first dose.
  Compound gossyrol acetate tablet: 20mg daily.

SUMMARY:
This is a single-arm, Phase II clinical study to explore the efficacy and safety of dalpiciclib combined with fluvestrant and compound gossypol acetate tablets in advanced HR-positive and HER2-negative breast cancer after CDK4/6 treatment failed.

DETAILED DESCRIPTION:
Dalpiciclib: According to the standard dose, 150mg orally for three weeks and stop for one week.

Fluvestrant: At the standard dose, 500mg once every four weeks. A further 500mg dose two weeks after the first dose.

Compound gossypol acetate tablets: 20mg once a day.

ELIGIBILITY:
Inclusion Criteria:

1.Written informed consent. 2.Women aged 18 years or older. 3.Eastern Cooperative Oncology Group(ECOG) has a physical fitness score of 0 or 1. 4.Life expectancy is more than six months. 5.Diagnosed as HR-positive HER2-negative metastatic breast cancer. 6.There was at least one measurable lesion according to RECIST 1.1. 7.Failed in treating with CDK4/6 inhibitors combined with endocrine therapy at the metastatic stage. 8.Good organ function. 9.Fertile female patients must have a negative serum pregnancy test within seven days prior to study treatment and consent to effective contraceptive use for 180 days from screening to the last dose of study treatment. 10.Female patients must agree not to breastfeed during the study period or for 180 days after the last dose of study therapy.

Exclusion Criteria:

1.Patients enrolled in any interventional clinical trial at the same time and received the investigational therapy ≤ four weeks prior to initiation of the regimen or at least five half-lives of the investigational drug. 2.Patients who had received radiation therapy with bone marrow coverage >20% within two weeks before the start of treatment, except for minor palliative radiation therapy more than one week before the first day of the study. 3.Patients with a visceral crisis, and requiring chemotherapy. 4.Patients allergic to dalpiciclib or compound gossyrol acetate tablets. 5.A history of platelet transfusion for chemotherapy-induced thrombocytopenia or prior cancer treatment (lasting > 4 weeks and associated with recent treatment) is known to result in ≥ grade 3 hematological toxicity. 6.The patient had any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML). 7.Patients have a severe, uncontrolled medical condition, a non-malignant systemic disease, or an active, uncontrolled infection. 8.Patients diagnosed, detected, or treated for another type of cancer within ≤2 years prior to beginning regimen therapy.

Patients with brain metastases or pial metastases uncontrolled. 9.Patients have received an allogeneic bone marrow transplant or double umbilical cord blood transplant. 10.Patients cannot swallow oral medications. 11.Patients with gastrointestinal disorders that may interfere with the absorption of investigational drugs. 12.Patients have had systemic active autoimmune disease (i.e., disease modulators, corticosteroids, or immunosuppressants) within the past two years. 13.Patients with a history of human immunodeficiency virus, active-hepatitis -B or C. 14.Pregnant or nursing women. Fertile adults without effective contraceptive methods.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  ORR is defined as the percentage of patients who achieved a best overall response of Complete Response (CR) or Partial Response (PR), per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions as assessed by the Investigator: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 24 months
  From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
Clinical Benefit Rate (CBR) | up to 24 months
  Percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) lasting 24 weeks or longer as defined in RECIST v1.1.
Duration of Overall Response(DoR) | up to 24 months
  Time from first recording to CR or PR to disease progression or all-cause death.
Time to response (TTR) | up to 24 months
  TTR defined as the time from the date of the first dose of study treatment to the first objective tumor response when CR or PR is observed.
Overall survival (OS) | up to 24 months
  Time to death from any cause from the date of first dose of study treatment
adverse event(AE) | Throughout the experiment, assessed up to 24 months.
  Evaluation performed using the National Cancer Institute (NCI)- Standard for Common Terminology for Adverse Events (CTCAE)v.5.0.

OTHER OUTCOMES:
Exploratory endpoint | Throughout the experiment, assessed up to 24 months.
  Correlation between the expression levels of LRPPRC and CDK6 and the efficacy of Dalpiciclib combined with Fulvestrant and Compound Gossyfol Acetate Tablets.

CONTACTS AND LOCATIONS:
Locations (1):
- zhejiangCH, Hangzhou, Zhejiang, China